CLINICAL TRIAL: NCT01294085
Title: Retrospective Analysis of the Difference of Prognosis Between Unresectable and Recurrent Biliary Tract Cancer
Brief Title: Case Series Study of Biliary Tract Cancer Patients in Japan
Status: Completed | Type: Observational
Sponsor: Kansai Hepatobiliary Oncology Group (Network)
Responsible Party: Sponsor
Other Study IDs: KHBO1001; UMIN000004530 (Registry Identifier: UMIN)
Record Dates: First submitted 2011-01-03; First posted 2011-02-11 (Estimated); Last update posted 2011-11-28 (Estimated); Status verified 2011-11

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To assess the difference of prognosis between unresectable and recurrent biliary tract cancer and evaluate prognostic factors.

DETAILED DESCRIPTION:
Most patients of biliary tract cancer have advanced disease at diagnosis and often relapse despite surgery. Combination therapy of gemcitabine and cisplatin could be a standard therapy for this kind of cancer with the evidence of phase III study compared with gemcitabine alone. However the prognosis and the tolerability of chemotherapy in the patients with recurrent biliary tract cancer after radical resection might differ from those of unresectable biliary tract cancer, because the dose intensity of chemotherapy can be influenced by adjuvant chemotherapy and/or hepatic resection.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable or recurrent biliary tract cancer

Exclusion Criteria:

* None

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
One year survival rate | 1 year

SECONDARY OUTCOMES:
Overall survival time | 3 years
Number of participants with adverse events | 3 years
Progression free survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuya Ioka, MD, Study Director — Osaka Medical Center for Cancer and CVD
Locations (1):
- Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka, Japan